CLINICAL TRIAL: NCT02176967
Title: Utilizing Response- and Biology-Based Risk Factors to Guide Therapy in Patients With Non-High-Risk Neuroblastoma
Brief Title: Response and Biology-Based Risk Factor-Guided Therapy in Treating Younger Patients With Non-high Risk Neuroblastoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL1232; NCI-2014-00677 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s15-00462; ANBL1232 (Other: Children's Oncology Group); ANBL1232 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Ganglioneuroblastoma; Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Neuroblastoma
MeSH Terms: conditions — Ganglioneuroblastoma; Neuroblastoma | interventions — Biopsy; Carboplatin; Watchful Waiting; Observation; Cyclophosphamide; Doxorubicin; Etoposide; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (clinical observation) (Experimental): Patients undergo clinical observation for 96 weeks in the absence of disease progression. Patients also undergo CT, MRI, and/or ultrasound throughout the trial.
  Interventions: Other: Clinical Observation; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound
- Group B (clinical observation, first-line chemotherapy) (Experimental): Patients undergo clinical observation for 3 years in the absence of disease progression. Upon disease progression, patients undergo surgery or receive first-line chemotherapy comprising carboplatin IV over 1 hour on day 1 (courses 1, 2, 4, 6, and 7), etoposide IV over 1 hour on days 1-3 (courses 1, 3, 4, 5, and 7), cyclophosphamide IV over 1 hour on day 1 (courses 2, 3, 5, 6, and 8), and doxorubicin hydrochloride IV over 15 minutes on day 1 (courses 2, 4, 6 and 8). Treatment with chemotherapy repeats every 21 days for 2-8 courses in the absence of disease progression or unacceptable toxicity. Once a PR or better is achieved, patients undergo clinical observation for 3 years. Patients also undergo CT, MRI, and/or ultrasound throughout the trial and undergo bone marrow aspiration, bone marrow biopsy, and tumor biopsy at screening and time of progression.
  Interventions: Procedure: Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Carboplatin; Other: Clinical Observation; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound
- Group C (clinical observation, first-line chemotherapy) (Experimental): Patients at high risk for deterioration and a poor outcome immediately receive first-line chemotherapy as in Group B. All other patients undergo clinical observation for 3 years in the absence of disease progression. Upon disease progression, patients receive first-line chemotherapy as in Group B. Once a PR or better is achieved, patients undergo clinical observation for 3 years. Patients also undergo CT, MRI, and/or ultrasound throughout the trial and undergo bone marrow aspiration, bone marrow biopsy, and tumor biopsy at screening and time of progression.
  Interventions: Procedure: Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Carboplatin; Other: Clinical Observation; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Other: Clinical Observation — Undergo clinical observation
  Other Names: observation
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Group B (clinical observation, first-line chemotherapy); Group C (clinical observation, first-line chemotherapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Ultrasound — Undergo ultrasound

SUMMARY:
This phase III trial studies how well response and biology-based risk factor-guided therapy works in treating younger patients with non-high risk neuroblastoma. Sometimes a tumor may not need treatment until it progresses. In this case, observation may be sufficient. Measuring biomarkers in tumor cells may help plan when effective treatment is necessary and what the best treatment is. Response and biology-based risk factor-guided therapy may be effective in treating patients with non-high risk neuroblastoma and may help to avoid some of the risks and side effects related to standard treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To eliminate therapy as the initial approach for infants < 12 months of age with small International Neuroblastoma Risk Group (INRG) stage L1 neuroblastoma while maintaining an overall survival (OS) of 99%.

II. To eliminate therapy as the initial approach for non-high-risk patients < 18 months of age with localized neuroblastoma and favorable biology (histologic and genomic features) while maintaining an OS of 99%.

III. To achieve a 3-year OS of > 81% for infants < 18 months of age with INRG stage Ms neuroblastoma using objective criteria for early initiation of a response-based treatment algorithm.

EXPLORATORY OBJECTIVES:

I. To describe the time to intervention or tumor progression, type of intervention and site of progression for patients with localized neuroblastoma who experience progression after an initial period of observation.

II. To characterize the pharmacokinetic profile of the chemotherapeutic agents carboplatin and etoposide in patients with stage Ms disease.

III. To define the genomic profile of tumors from patients with non-high-risk neuroblastoma both at initial biopsy and at the time of subsequent biopsy or surgical resection.

IV. To describe the histology of tumor specimens obtained at the time of subsequent biopsy or surgical resection.

V. To determine the salvage rate (OS) of patients with tumor relapse or disease progression.

VI. To determine the procedural complication rate (initial biopsy, resection [intraoperative and postoperative], subsequent biopsy) and correlate with the degree of surgical resection.

VII. To determine the rate of reduction in image defined risk factors (IDRF) in L2 tumors following observation or chemotherapy.

OUTLINE: Patients are assigned to 1 of 3 treatment groups.

GROUP A: Patients undergo clinical observation for 96 weeks in the absence disease progression. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), and/or ultrasound throughout the trial.

GROUP B: Patients undergo clinical observation for 3 years in the absence of disease progression. Upon disease progression, patients undergo surgery or receive first-line chemotherapy comprising carboplatin intravenously (IV) over 1 hour on day 1 (courses 1, 2, 4, 6, and 7), etoposide IV over 1 hour on days 1-3 (courses 1, 3, 4, 5, and 7), cyclophosphamide IV over 1 hour on day 1 (courses 2, 3, 5, 6, and 8), and doxorubicin hydrochloride IV over 15 minutes on day 1 (courses 2, 4, 6 and 8). Treatment with chemotherapy repeats every 21 days for 2-8 courses in the absence of disease progression or unacceptable toxicity. Once a partial response (PR) or better is achieved, patients undergo clinical observation for 3 years. Patients also undergo CT, MRI, and/or ultrasound throughout the trial and undergo bone marrow aspiration, bone marrow biopsy, and tumor biopsy at screening and time of progression.

GROUP C: Patients at high risk for deterioration and a poor outcome immediately receive first-line chemotherapy as in Group B. All other patients undergo clinical observation for 3 years in the absence of disease progression. Upon disease progression, patients receive first-line chemotherapy as in Group B. Once a PR or better is achieved, patients undergo clinical observation for 3 years. Patients also undergo CT, MRI, and/or ultrasound throughout the trial and undergo bone marrow aspiration, bone marrow biopsy, and tumor biopsy at screening and time of progression.

After completion of study treatment, patients are followed up annually for up to 10 years post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be:

  * < 12 months (< 365 days) of age at diagnosis with INRG stage L1; or
  * < 18 months (< 547 days) of age at diagnosis with INRG stage L2 or stage Ms neuroblastoma/ganglioneuroblastoma
* Enrollment on ANBL00B1 or APEC14B1 is required for all newly diagnosed patients
* Patients must have newly diagnosed v-myc avian myelocytomatosis viral oncogene neuroblastoma derived homolog (MYCN) non-amplified neuroblastoma (International Classification of Diseases for Oncology [ICD-O] morphology 9500/3) or MYCN non-amplified ganglioneuroblastoma verified by histology
* Patients must meet the specified criteria for one of the treatment groups defined below; genomic features include MYCN gene amplification, segmental chromosome aberrations (somatic copy number loss at 1p, 3p, 4p, or 11q or somatic copy number gain at 1q, 2p, or 17q) and deoxyribonucleic acid (DNA) index

  * "Favorable" genomic features are defined by one or more whole-chromosome gains or hyperdiploid tumor (DNA index > 1) in the absence of segmental chromosome aberrations as defined above
  * "Unfavorable" genomic features are defined by the presence of any segmental chromosome aberration (somatic copy number loss at 1p, 3p, 4p, or 11q or somatic copy number gain at 1q, 2p, or 17q) or diploid tumor (DNA index = 1); this includes copy neutral loss of heterozygosity (LOH)
  * Only patients with MYCN non-amplified tumors are eligible for this study
* Group A: patients < 12 months (< 365 days) of age with newly diagnosed INRG stage L1 neuroblastoma/ganglioneuroblastoma who meet the following criteria:

  * Greatest tumor diameter < 5 cm of adrenal or non-adrenal origin
  * Patients with non-adrenal primaries are eligible, but must have positive uptake on metaiodobenzylguanidine (MIBG) scan or elevated catecholamine metabolites (urine or serum) to support the diagnosis of neuroblastoma
  * No prior tumor resection or biopsy
* Group A will be further split into two subsets, which are mutually exclusive, for statistical purposes

  * Group A1:

    * > 6 months and < 12 months of age with an adrenal primary tumor < 5 cm in greatest diameter OR
    * Patients less than 6 months of age with an adrenal primary tumor > 3.1 and < 5 cm in greatest diameter OR
    * < 12 months of age with a non-adrenal primary site < 5 cm in greatest diameter
  * Group A2: =< 6 months of age with an adrenal primary site and tumor =< 3.1 cm in greatest diameter
* Group B: patients < 18 months (< 547 days) of age with newly diagnosed INRG stage L2 neuroblastoma/ganglioneuroblastoma who meet the following criteria:

  * No life threatening symptoms or no impending neurologic or other organ function compromise (e.g. epidural or intraspinal tumors with existing or impending neurologic impairment, periorbital or calvarial-based lesions with existing or impending cranial nerve impairment, anatomic or mechanical compromise of critical organ function by tumor [abdominal compartment syndrome, urinary obstruction, etc.]); horner syndrome is not considered neurologic compromise
  * No prior tumor resection, tumor biopsy ONLY
  * Only patients with both favorable histology and favorable genomic features will remain on study as part of Group B; the institution will be notified of histologic and genomic results within 3 weeks of specimen submission on ANBL00B1 or APEC14B1
* Group C: patients < 18 months (< 547 days) of age with newly diagnosed INRG stage Ms neuroblastoma/ganglioneuroblastoma
* No prior radiotherapy or chemotherapy, with the exception of dexamethasone, which is allowed
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with MYCN amplified tumors are not eligible
* Group B and C patients who do not enroll on ANBL1232 within 4 weeks of definitive diagnostic procedure
* Group A and C patients, not required to undergo tumor biopsy, who do not enroll on ANBL1232 within 4 weeks of confirmatory imaging study

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 621 (Estimated)
Dates: Start 2014-08-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) (Strata 1-4) | From date of enrollment until death or last contact, assessed up to 3 years
  The Kaplan-Meier method will be used to estimate the 3-year overall survival for each stratum. OS is measured from time of enrollment to the date of death from any cause.

OTHER OUTCOMES:
Time to intervention or tumor progression | Up to 3 years
  Will be assessed by a descriptive analysis for the cohort of patients with localized tumors who progress after an initial period of observation.
Type of intervention required | Up to 3 years
  Will be assessed by a descriptive analysis for the cohort of patients with localized tumors who progress after an initial period of observation.
Site of progression | Up to 3 years
  Will be assessed by a descriptive analysis for the cohort of patients with localized tumors who progress after an initial period of observation.
Pharmacokinetic (PK) profile of carboplatin and etoposide in patients with stage Ms disease, including peak concentration, area under the curve, clearance, volume of distribution, half-life, and mean residence time | Pre-dose, 1, 2, 4, 8, and 24 hours on days 1 and 2 of either course 1 or 7
  The coefficient of variation will be calculated to quantify the degree of inter-patient and intra-patient variability of etoposide and carboplatin PK. The relationship between patient characteristics will be assessed graphically in an exploratory fashion and with regression models and if appropriate, Spearman's rank correlation coefficient will be used. Correlations between PK parameters and the symptom score and hepatic and renal dysfunction will be explored. Logistic regression models adjusting for patient level covariates will be explored.
Genomic profile of tumors | Up to time of biopsy or surgical resection
  Will be assessed by determining the presence or absence of each segmental aberration (segmental loss at 1p, 3p, 4p, or 11q or segmental gain at 1p, 2p, or 17q), both at initial biopsy and at the time of subsequent biopsy or surgical resection, and correlating with patient characteristics using a chi-squared test and with outcome using a log-rank test. In cases with specimens from diagnosis and at the time of subsequent biopsy/resection, the profiles will be compared focusing on changes in the copy number pattern.
Histology of tumor specimens | Up to time of biopsy or surgical resection
  Will be assessed by a descriptive analysis of the histology of tumor specimens obtained at the time of subsequent biopsy or surgical resection.
Salvage rate (overall survival [OS]) of patients with tumor relapse or disease progression | From the date of enrollment until death or until last contact if the patient is alive, assessed up to 3 years
  Will be assessed by calculating the overall survival for the cohort of patients with tumor relapse or disease progression.
Procedural complication rate | Up to 60 days after surgery
  Will be assessed by determining the complication rate for each type of procedure (initial biopsy and resection [intraoperative and postoperative]) and correlating the occurrence of surgical complications with the degree of surgical resection using a Wilcoxon rank-sum test (to account for the ordering of the surgical resection categories).
Rate of reduction in Image Defined Risk Factors (IDRF) in L2 tumors | Up to 3 years
  Will be assessed by computing the proportion of patients with L2 tumors for which each particular IDRF and any IDRF is present at diagnosis and then absent after observation or chemotherapy. In addition, McNemar's test for paired observations will be applied to determine whether there is a difference in the proportion of each IDRF and any IDRF present before and after observation or chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Holly J Meany, Principal Investigator — Children's Oncology Group
Locations (222):
- United States (193):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (17):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Jim Pattison Children's Hospital, Saskatoon, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia